CLINICAL TRIAL: NCT03251963
Title: Fixed Versus Weight-Based Enoxaparin Dosing in Thoracic Surgery Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Principal Investigator, Christopher Pannucci, Assistant Professor, University of Utah
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 100484
Record Dates: First submitted 2017-08-14; First posted 2017-08-16 (Actual); Results first posted 2020-07-08 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Venous Thromboembolism; Deep Venous Thrombosis; Surgery
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis | interventions — Enoxaparin

STUDY DESIGN:
Intervention Model Description: Participants enrolled in months 1-6 of the study will all receive a fixed dose of enoxaparin. Patients enrolled in months 7-12 of the study will all receive a variable dose of enoxaparin.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Fixed Dose Enoxaparin (Experimental): Eligible patients will be administered 40 mg enoxaparin daily and will have steady state peak and trough anti-Xa levels drawn after the third enoxaparin dose.
  Interventions: Drug: Fixed Dose Enoxaparin
- Variable Dose Enoxaparin (Experimental): Eligible patients will be administered 0.5 mg/kg enoxaparin daily and will have steady state peak and trough anti-Xa levels drawn after the third enoxaparin dose.
  Interventions: Drug: Variable Dose Enoxaparin

INTERVENTIONS:
Drug: Fixed Dose Enoxaparin — Eligible patients will be administered 40 mg enoxaparin daily and will have steady state peak and trough anti-Xa levels drawn after the third enoxaparin dose. For patients in-range (levels 0.3-0.5IUmL), no intervention will be undertaken. For patients out of range, enoxaparin dose will be adjusted according to an established dose adjustment algorithm. Repeat levels will be checked after the third administration of the new dose.
  Arms: Fixed Dose Enoxaparin
Drug: Variable Dose Enoxaparin — Eligible patients will be administered 0.5 mg/kg enoxaparin daily and will have steady state peak and trough anti-Xa levels drawn after the third enoxaparin dose. For patients in-range (levels 0.3-0.5IUmL), no intervention will be undertaken. For patients out of range, enoxaparin dose will be adjusted according to an established dose adjustment algorithm. Repeat levels will be checked after the third administration of the new dose.
  Arms: Variable Dose Enoxaparin

SUMMARY:
The aim of this research is to better understand how patient-level factors can be used to predict the appropriate enoxaparin dose to maximize venous thromboembolism (VTE) risk reduction and minimize bleeding.

DETAILED DESCRIPTION:
VTE encompasses deep venous thrombosis and pulmonary embolus and is the proximate cause of death in over 100,000 hospitalized patients per year 4,5. To put this in better context, VTE kills more people each year than the annual morbidity from motor vehicle crashes and breast cancer combined-and one third of these deaths are known to occur after surgical procedures 34. "Breakthrough" VTE events occur in patients despite the receipt of guideline-compliant chemical prophylaxis. These events can be frustrating for surgeons, can represent a resource and financial burden for hospital systems, and most importantly, can be life or limb threatening for patients.

Existing data from our group and others suggests that inadequate enoxaparin dosing, quantified by aFXa levels, represents a plausible explanatory mechanism for "breakthrough" VTE events that occur among thoracic surgery patients. This project will examine the pharmacodynamics of fixed dose enoxaparin (40mg/day) after VATS-this dose and frequency were the most commonly prescribed VTE chemical prophylaxis strategy in a recent survey of thoracic surgeons 35. If inadequate aFXa levels are observed with fixed enoxaparin dosing, the study will design, implement and test a weight-based dosing approach to optimize aFXa levels. The study will also examine how alteration of enoxaparin dose magnitude affects peak aFXa levels and risk for VTE and major bleeding events.

Aim 1: To evaluate peak steady-state aFXa levels in response to a fixed dose of enoxaparin prophylaxis (40mg once daily) in VATS patients.

Rationale: Over 12% of thoracic surgery patients have "breakthrough" VTE events despite receipt of fixed dose chemical prophylaxis 29. Fixed dose enoxaparin prophylaxis has been shown to be inadequate for the majority of patients in other surgical subspecialties.

Hypothesis: Peak steady state aFXa levels will be within the accepted range (0.3-0.5 IU/mL) in 40% of patients after VATS.

Aim 2: To compare the effect of fixed (40mg once daily) and weight-based (0.5mg/kg once daily) enoxaparin prophylaxis on peak steady state aFXa levels after VATS.

Rationale: Our preliminary data shows a potential association between body weight and aFXa levels in response to fixed dosing; this will be confirmed using a multi-center approach in Aim #1. Body weight may be an important predictor of appropriate enoxaparin dose.

Hypothesis: Weight-based enoxaparin prophylaxis, when compared to fixed dose prophylaxis, will increase the proportion of patients with in-range peak aFXa levels from 40% to 80%.

Aim 3: To examine rates of 90-day VTE and clinically relevant bleeding events in VATS patients who receive fixed dose vs. weight-based enoxaparin prophylaxis.

Rationale: This observational Aim will allow us to better understand VTE and bleeding rates after VATS. Since these are rare events it is impossible to power the study to detect increases or decreases in risk between the dose groups. This study does provide a way to demonstrate an unexpected, very large difference in risk.

Hypothesis: Rates of post-operative VTE and clinically relevant bleeding will be less than 2% in each group.

ELIGIBILITY:
Inclusion Criteria:

* receiving Video-Assisted Thoracoscopic Surgery
* able to have Enoxaparin initiated within 8 hours after procedure

Exclusion Criteria:

* Contraindication to use of enoxaparin
* Intracranial bleeding/stroke
* Hematoma or bleeding disorder
* Heparin-induced thrombocytopenia positive
* Creatinine clearance less than or equal to 30 mL/min
* Serum creatinine greater than 1.6 mg/dL
* Epidural catheter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2019-03-27 (Actual); Study Completion 2019-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Puccini, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Pannucci CJ, Fleming KI, Varghese TK Jr, Stringham J, Huang LC, Pickron TB, Prazak AM, Bertolaccini C, Momeni A. Low Anti-Factor Xa Level Predicts 90-Day Symptomatic Venous Thromboembolism in Surgical Patients Receiving Enoxaparin Prophylaxis: A Pooled Analysis of Eight Clinical Trials. Ann Surg. 2022 Dec 1;276(6):e682-e690. doi: 10.1097/SLA.0000000000004589. Epub 2020 Oct 19. PMID 33086312
- [Derived] Pannucci CJ, Fleming KI, Bertolaccini C, Moulton L, Stringham J, Barnett S, Lin J, Varghese TK Jr. Fixed or Weight-Tiered Enoxaparin After Thoracic Surgery for Venous Thromboembolism Prevention. Ann Thorac Surg. 2020 Jun;109(6):1713-1721. doi: 10.1016/j.athoracsur.2019.12.058. Epub 2020 Feb 8. PMID 32045583

RESULTS

PARTICIPANT FLOW:
Groups:
- Weight Tiered Enoxaparin: Eligible patients will be receive weight tiered daily enoxaparin. Patients <70kg received 30mg, patients 70kg to 89.9kg received 40mg, and patients ≥90kg received 50mg.
  Variable Dose Enoxaparin: Patients <70kg received 30mg, patients 70kg to 89.9kg received 40mg, and patients ≥90kg received 50mg. For patients in-range (levels 0.3-0.5IUmL), no intervention will be undertaken. For patients out of range, enoxaparin dose will be adjusted according to an established dose adjustment algorithm. Repeat levels will be checked after the third administration of the new dose.
Period: Overall Study
Arm/Group | Fixed Dose Enoxaparin | Weight Tiered Enoxaparin
Started | 65 | 66
Completed | 56 | 61
Not Completed | 9 | 5
Not completed — inappropriate Xa level timing | 6 | 3
Not completed — no peak Xa level drawn | 2 | 0
Not completed — bled prior to Xa level | 1 | 2

BASELINE CHARACTERISTICS:
Population: Group 1 65 plus Group 2 66 =131 total
Groups:
- Total: Total of all reporting groups
Arm/Group | Fixed Dose Enoxaparin | Weight Tiered Enoxaparin | Total
Number analyzed (Participants) | 65 | 66 | 131
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 33 | 65
  >=65 years | 33 | 33 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (15.6) | 59.0 (16.8) | 60.0 (16.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 32 | 69
  Male | 28 | 34 | 62
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 1 | 0 | 1
  White | 61 | 63 | 124
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 65 | 66 | 131

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With in Range Initial Peak Xa Level
Description: Number of patients with in range initial peak Xa level
Time Frame: 36 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Fixed Dose Enoxaparin | Weight Tiered Enoxaparin
Number analyzed (Participants) | 56 | 61
Participants | 27 | 27

2. Secondary Outcome: Number of Participants With Venous Thromboembolism Events or Death
Description: Any symptomatic venous thromboembolism events, including deep venous thrombosis or pulmonary embolus occurring within 90 days of surgery
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Fixed Dose Enoxaparin | Weight Tiered Enoxaparin
Number analyzed (Participants) | 65 | 66
Participants | 1 | 0

3. Secondary Outcome: Number of Participants With Bleeding Events
Description: Bleeding events requiring alteration in the course of care within 90 days of surgery
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Fixed Dose Enoxaparin | Weight Tiered Enoxaparin
Number analyzed (Participants) | 65 | 66
Participants | 1 | 3

ADVERSE EVENTS:
Time Frame: 90 days
Description: Symptomatic VTE was defined as any symptomatic deep vein thrombosis or pulmonary embolus with imaging confirmation. Screening duplex ultrasound was not performed, as suggested by current American College of Chest Physicians guidelines. Clinically relevant bleeding was defined as any bleeding that changed the course of care; this included bleeding requiring enoxaparin cessation, unexpected transfusion, or procedural (interventional radiology or operating room) intervention.
Arm/Group | Fixed Dose Enoxaparin | Weight Tiered Enoxaparin
All-Cause Mortality (participants affected / at risk) | 1/65 | 0/66
Serious Adverse Events (participants affected / at risk) | 1/65 | 0/66
Other Adverse Events (participants affected / at risk) | 1/65 | 3/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fixed Dose Enoxaparin (N=65) | Weight Tiered Enoxaparin (N=66)
90-day Death (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fixed Dose Enoxaparin (N=65) | Weight Tiered Enoxaparin (N=66)
DVT/PE (Blood and lymphatic system disorders) | 0 | 0 — 90 day symptomatic VTE
clinically relevant bleeding (Blood and lymphatic system disorders) | 1 | 3 — 90-day clinically relevant bleeding

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-19): https://cdn.clinicaltrials.gov/large-docs/63/NCT03251963/Prot_SAP_001.pdf